CLINICAL TRIAL: NCT02443805
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Study of the Efficacy and Safety of STG320 Sublingual Tablets of House Dust Mite (HDM) Allergen Extracts in Adults and Adolescents With HDM-associated Allergic Rhinitis
Brief Title: Efficacy & Safety of STG320 Sublingual Tablets of HDM Allergen Extracts in Adults and Adolescents With HDM-associated AR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SL75.14
Record Dates: First submitted 2015-04-29; First posted 2015-05-14 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-09

CONDITIONS: Rhinitis, Allergic, Perennial; House Dust Mite Allergy
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Dust Mite Allergy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 300 IR (Active Comparator): 300 IR tablet of HDM Allergen Extracts
  Interventions: Biological: 300 IR
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: 300 IR — 300 IR tablet of HDM Allergen Extracts
  Arms: 300 IR
Biological: Placebo — Placebo tablet
  Arms: Placebo

SUMMARY:
The objective of this study was to assess the efficacy and safety of 12 months of treatment with 300 IR of STG320 sublingual tablets compared with placebo in adults and adolescents with HDM-associated allergic rhinitis.

DETAILED DESCRIPTION:
This study was a randomized, double-blind, placebo-controlled, phase III study with 2 parallel arms in adults and adolescents with HDM-associated allergic rhinitis (AR) for at least one year.

The primary objective was to assess the efficacy of STG320 sublingual tablets at a daily dosage of 300 IR when administered for 12 months to adults and adolescents with HDM-associated AR. The primary efficacy variable was the average Total Combined Score.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients with HDM-associated allergic rhinitis (AR) for at least 1 year
* Patients sensitized to D. pteronyssinus (D. pte) and/or D. farinae (D. far) defined on skin prick test and HDM-specific serum IgE

Main Exclusion Criteria:

* A history of rhinitis, rhinoconjunctivitis or asthma to allergens other than HDM, likely to result in rhinitis symptoms during the evaluation periods
* Partly controlled or uncontrolled asthma
* Controlled asthma requiring controller treatment(s) consistent with GINA 2014 treatment Steps 3 to 5

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1607 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Demoly, MD, Principal Investigator — CHU Arnaud de Villeneuve, Montpellier, France; Tom Casale, MD, Principal Investigator — University of South of Florida, Tampa, USA
Locations (2):
- University of South of Florida, Tampa, Florida, United States
- CHU Arnaud de Villeneuve, Montpellier, France

REFERENCES:
- [Derived] Worm M, Demoly P, Okamoto Y, Vidal C, Daghildjian K, Yan K, Casale TB, Bergmann KC. Safety of 300IR house dust mite sublingual tablet from pooled clinical trial and post-marketing data. World Allergy Organ J. 2024 Jun 25;17(7):100924. doi: 10.1016/j.waojou.2024.100924. eCollection 2024 Jul. PMID 39035788
- [Derived] Pfaar O, De Blay F, Canonica GW, Casale TB, Gevaert P, Hellings PW, Kowal K, Passalacqua G, Tortajada-Girbes M, Vidal C, Worm M, Bahbah F, Demoly P. Clinical benefits with 300 IR HDM SLIT tablet in Europeans with house dust mite allergic rhinitis: Post hoc analysis of a large phase 3 trial. World Allergy Organ J. 2023 Dec 22;17(1):100849. doi: 10.1016/j.waojou.2023.100849. eCollection 2024 Jan. PMID 38225952

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between 29 September 2015 (first patient, first visit) and 25 June 2018 (last patient, last visit).
Pre-assignment Details: 2,174 (50.9%) and 486 (11.4%) patients were excluded before and during the placebo run-in period, respectively. The main reason for screen failures at these two stages was a failure to meet randomization criteria.
Period: Overall Study
Arm/Group | 300 IR | Placebo
Started | 802 | 805
Completed | 589 | 678
Not Completed | 213 | 127
Not completed — Adverse Event | 100 | 18
Not completed — Withdrawal by Subject | 73 | 74
Not completed — Lost to Follow-up | 19 | 14
Not completed — Pregnancy | 6 | 5
Not completed — Protocol Violation | 2 | 4
Not completed — Lack of Efficacy | 1 | 1
Not completed — Non-compliance with study drug | 6 | 4
Not completed — Withdrawal by parent/guardian | 3 | 5
Not completed — Any other reason not above-mentioned | 3 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all randomized patients who received at least one dose of the IP of treatment period and had at least one primary efficacy evaluation during the overall treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | 300 IR | Placebo | Total
Number analyzed (Participants) | 711 | 765 | 1476
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (13.07) | 29.6 (12.58) | 29.6 (12.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 360 | 396 | 756
  Male | 351 | 369 | 720
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 46 | 96
  Not Hispanic or Latino | 660 | 719 | 1379
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 21 | 20 | 41
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 25 | 37 | 62
  White | 660 | 701 | 1361
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  North America | 212 | 240 | 452
  Europe | 453 | 477 | 930
  Israel | 23 | 23 | 46
  Russia | 23 | 25 | 48

OUTCOME MEASURES:

1. Primary Outcome: Total Combined Score
Description: Average Total Combined Score (TCS), calculated for each patient as the average of the non-missing daily TCSs during the primary evaluation period. The daily TCS (scale 0-15) was the sum of the patient's daily Rhinitis Total Symptom Score (RTSS, scale 0-12) and daily Rescue Medication Score (RMS, scale 0-3). Lower is better.
Time Frame: 12 months
Population: The FAS included all randomized patients (pts) who received at least one dose of the IP of treatment period and had at least one primary efficacy evaluation during the overall treatment period: 1,476 pts. Among these pts, only those with efficacy evaluation during the primary evaluation period were included in the primary analysis: 1,262 pts.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | 300 IR | Placebo
Number analyzed (Participants) | 586 | 676
Units on a scale | 3.62 [3.33 to 3.92] | 4.35 [4.06 to 4.66]
Statistical Analysis 1: Comparison: 300 IR vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — Source Model: Type III effects Covariates: Treatment group, Gender, Age Class, Sensitization Status, Asthma Status, Pooled Center, Baseline Average RTSS

2. Secondary Outcome: Average Rhinitis Total Symptom Score (RTSS)
Description: Average RTSS during the primary evaluation period. The daily Total Symptom Scores (RTSS) was the sum of the 4 rhinitis symptom scores: sneezing, rhinorrhoea, nasal pruritus and nasal congestion, each graded on a 4-point scale (0-3; 0: absent, 1: mild, 2: moderate, 3: severe).
  It ranges from 0 to 12. Lower is better.
Time Frame: 12 months
Population: The FAS included all randomized patients (pts) who received at least one dose of the IP of treatment period and had at least one primary efficacy evaluation during the overall treatment period: 1,476 pts. Among these pts, only those with efficacy evaluation during the primary evaluation period were included in the secondary analysis: 1,262 pts.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | 300 IR | Placebo
Number analyzed (Participants) | 586 | 676
Units on a scale | 3.16 [2.89 to 3.43] | 3.79 [3.53 to 4.07]

3. Secondary Outcome: Average Rescue Medication Score (RMS)
Description: Average RMS during the primary evaluation period. Rescue Medication Score (RMS) ; range 0-3, lower is better.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | 300 IR | Placebo
Number analyzed (Participants) | 586 | 676
Units on a scale | 0.21 [0.17 to 0.25] | 0.30 [0.26 to 0.35]

ADVERSE EVENTS:
Time Frame: 12 months
Description: Safety variables were adverse events (AEs) monitored throughout the study and data from physical examinations and clinical laboratory assessments.
  1,607 patients were randomized. 6 patients randomized by mistake did not receive any IP of the treatment period and were excluded from the Safety Set.
  Accordingly, the Safety Set comprised 1,601 patients.
Arm/Group | 300 IR | Placebo
All-Cause Mortality (participants affected / at risk) | 0/800 | 0/801
Serious Adverse Events (participants affected / at risk) | 21/800 | 9/801
Other Adverse Events (participants affected / at risk) | 424/800 | 223/801
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 300 IR (N=800) | Placebo (N=801)
Appendicitis (Infections and infestations) | 3 | 0
Tick-borne viral encephalitis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 | 0
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1 | 0
Plica syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Chronic fatigue syndrome (General disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 300 IR (N=800) | Placebo (N=801)
Oral pruritus (Gastrointestinal disorders) | 189 | 29
Oedema mouth (Gastrointestinal disorders) | 112 | 3
Tongue oedema (Gastrointestinal disorders) | 68 | 3
Lip oedema (Gastrointestinal disorders) | 61 | 8
Dysphagia (Gastrointestinal disorders) | 53 | 2
Nausea (Gastrointestinal disorders) | 47 | 8
Abdominal pain upper (Gastrointestinal disorders) | 43 | 12
Nasopharyngitis (Infections and infestations) | 107 | 117
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 136 | 27
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 46 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 45 | 31
Ear pruritus (Ear and labyrinth disorders) | 115 | 13
Headache (Nervous system disorders) | 57 | 68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT02443805/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT02443805/SAP_001.pdf